CLINICAL TRIAL: NCT01341275
Title: Project to Evaluate Hepatitis B Vaccine-induced Immunity Among US-born Adolescents Who Received Hepatitis B Primary Vaccination Series During Early Childhood
Brief Title: Adolescents' Response to Hepatitis B Vaccine Booster Dose
Acronym: REACH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Amy B. Middleman, MD, MSEd, MPH/Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-26257
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Hepatitis B
Keywords: hepatitis B vaccine; duration of protection; adolescent immunization; anamnestic response; booster dose; Immunity to hepatitis B as measured by anti-HBSAg titers
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- birth, lower dose booster (Experimental): Adolescents who received their first dose of hepatitis B vaccine at or before day 7 of life who received a 10 ug dose of hepatitis B vaccine as a booster
  Interventions: Biological: hepatitis B vaccine
- birth, higher dose booster (Experimental): Adolescents who received their first dose of hepatitis B vaccine at or before day 7 of life who received a 20 ug dose of hepatitis B vaccine as a booster
  Interventions: Biological: hepatitis B vaccine
- 4 weeks, lower dose booster (Experimental): Adolescents who received their first dose of hepatitis B vaccine at or after 4 weeks of life who received a 10 ug dose of hepatitis B vaccine as a booster
  Interventions: Biological: hepatitis B vaccine
- 4 weeks, higher dose booster (Experimental): Adolescents who received their first dose of hepatitis B vaccine at or after 4 weeks of life who received a 20 ug dose of hepatitis B vaccine as a booster
  Interventions: Biological: hepatitis B vaccine

INTERVENTIONS:
Biological: hepatitis B vaccine — 10 ug dose, one-time administration
  Other Names: EngerixB
  Arms: 4 weeks, lower dose booster; birth, lower dose booster
Biological: hepatitis B vaccine — 20 ug dose, one-time administration
  Other Names: EngerixB
  Arms: 4 weeks, higher dose booster; birth, higher dose booster

SUMMARY:
The aims of this study are to determine:

1. the degree of immunity against hepatitis B,
2. factors associated with immunity against hepatitis B,
3. if the amount of antigen provided in a booster dose (used to measure the degree of immune memory) affects the body's response to the booster, and
4. if the age at which the vaccination was initiated during infancy affects duration of protection against hepatitis B among adolescents 16-19 years of age born in the United States who were immunized against hepatitis B as infants. These data will be important to evaluate the potential need for a possible booster dose of hepatitis B vaccine among adolescents.

Study subjects eligible for enrollment will:

* have blood drawn for baseline serologies
* receive the hepatitis B booster dose (randomly determined to be either a 10 ug or 20 ug dose)
* have blood drawn again 14 days later to determine if the booster dose has engendered an anamnestic response (a response attributed to prior immunity rather than a new response to the vaccine)

The primary hypothesis is that the majority of young people will exhibit immune memory for hepatitis B in response to a booster dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 16-19 years of age
* born in the United States
* received the full hepatitis B vaccination series by 12 months of age
* received the third dose of hepatitis B vaccine within 10 months of the first dose

Exclusion Criteria:

* a history of hepatitis B disease
* being born to a mother with hepatitis B at the time of the participant's birth
* having received hepatitis B immune globulin as an infant
* immunosuppression including HIV or chronic/current steroid use (use > 10 days duration within the 3 months of enrollment)
* renal insufficiency or dialysis
* pregnancy (due to theoretical risk of different immune response among pregnant females)
* ever receiving a booster (fourth) dose of hepatitis B vaccine
* history of allergy to the hepatitis B vaccine
* receipt of blood products or IgG within 3 months of enrollment
* having received another vaccine within 2 weeks of enrollment

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
anti-HBSAg titers | 13-15 days after enrollment and booster dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - Texas Children's Pediatric Associates, Houston, Texas

REFERENCES:
- [Derived] Spradling PR, Kamili S, Xing J, Drobeniuc J, Hu DJ, Middleman AB. Response to challenge dose among young adults vaccinated for hepatitis B as infants: importance of detectable residual antibody to hepatitis B surface antigen. Infect Control Hosp Epidemiol. 2015 May;36(5):529-33. doi: 10.1017/ice.2015.6. Epub 2015 Feb 3. PMID 25643863
- [Derived] Middleman AB, Baker CJ, Kozinetz CA, Kamili S, Nguyen C, Hu DJ, Spradling PR. Duration of protection after infant hepatitis B vaccination series. Pediatrics. 2014 Jun;133(6):e1500-7. doi: 10.1542/peds.2013-2940. Epub 2014 May 19. PMID 24843060